CLINICAL TRIAL: NCT04605133
Title: Electrical Impedance Tomography Monitoring and Invasive Mechanical Ventilation During Pronation in Acute Respiratory Distress Syndrome.
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Azienda Sanitaria-Universitaria Integrata di Udine (Other)
Responsible Party: Principal Investigator, Luigi Vetrugno, Clinical Professor in Anesthesiology and Intensive Care, Azienda Sanitaria-Universitaria Integrata di Udine
Other Study IDs: EIT during pronation in ARDS
Record Dates: First submitted 2020-10-06; First posted 2020-10-27 (Actual); Last update posted 2021-07-21 (Actual); Status verified 2021-07

CONDITIONS: ARDS, Human
MeSH Terms: conditions — Respiratory Distress Syndrome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- ARDS: Patients with mild or severe ARDS necessitating of prone position during mechanical ventilation
  Interventions: Device: Electrical impedance tomography

INTERVENTIONS:
Device: Electrical impedance tomography — Every patient is monitored with electrical impedance tomograpy before, during and after prone position.

SUMMARY:
Acute respiratory distress syndrome is an acute form of lung injury. The most commonly used classification criteria for this syndrome are Berlin's Criteria. The actual literature underlines the advantages of prone position in mild or severe forms of ARDS in association with invasive mechanical ventilation. The hypothesis of this study is to investigate the effective ventilation and perfusion modifications during pronation assessed with clinical parameters and with the aid of the electrical impedance tomography.

ELIGIBILITY:
Inclusion Criteria:

* mild or severe ARDS according to Berlin's Criteria
* recruitment maximum 72 hours from the diagnosis of ARDS

Exclusion Criteria:

* other non-ARDS respiratory system pathologies
* hemodynamic instability (mean arterial pressure < 60 mmHg)
* pneumothorax
* endocranial hypertension
* skin lesions or burns
* presence of pacemaker or implantable defibrillator
* pregnancy

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients' anthropometric data were collected. Ventilation parameters, electric impedence tomography parameters and blood gas analysis values were collected four times: patient supine (T0), one hour after pronation (T1), sixteen hours after pronation (T2), one hour after supination (T3).
Sampling Method: Non-Probability Sample
Enrollment: 15 (Estimated)
Dates: Start 2020-06-01 (Actual); Primary Completion 2020-12-31 (Actual); Study Completion 2021-12-31 (Estimated)

PRIMARY OUTCOMES:
Pronation and Regions of Interest increase in percentage | 1 hour after supination
  Demonstrate that pronation, without any recruitment maneuver, augments the dorsal regions of interest of 5%.

SECONDARY OUTCOMES:
PaO2/FiO2 ratio and ventral/dorsal Regions of Interest ratio | 1 hour after supination
  Obtain a statistical significant increase of PaO2/FiO2 ratio, with a consensual decrease of the ventral/dorsal Region of Interest ratio. It'a a measure of the difference between two ratios.
Homogeneity of the ventral and dorsal regions from 0 to 1 | 1 hour after supination
  Verify in which of the 4 measurements (T0-T1-T2-T3) the ventral/dorsal Region of Interest ratio is closer to 1, which means a complete homogeneity of the ventral and dorsal regions.
Region of Interest ratio and days of mechanical ventilation. | 30 days after pronation
  Understand if there is an association between ROI ratio and the days of mechanical ventilation.
Region of Interest ratio and length of stay in intensive care unit | 30 days after pronation
  Understand if there is an association between ROI ratio and the length of stay in intensive care unit.

CONTACTS AND LOCATIONS:
Locations (1):
- Anesthesiology and Intensive Care Clinic - Department of Medicine - ASUIUD, Udine, Italy

REFERENCES:
- [Background] ARDS Definition Task Force; Ranieri VM, Rubenfeld GD, Thompson BT, Ferguson ND, Caldwell E, Fan E, Camporota L, Slutsky AS. Acute respiratory distress syndrome: the Berlin Definition. JAMA. 2012 Jun 20;307(23):2526-33. doi: 10.1001/jama.2012.5669. PMID 22797452
- [Background] Mauri T, Eronia N, Abbruzzese C, Marcolin R, Coppadoro A, Spadaro S, Patroniti N, Bellani G, Pesenti A. Effects of Sigh on Regional Lung Strain and Ventilation Heterogeneity in Acute Respiratory Failure Patients Undergoing Assisted Mechanical Ventilation. Crit Care Med. 2015 Sep;43(9):1823-31. doi: 10.1097/CCM.0000000000001083. PMID 25985386
- [Background] Cinnella G, Grasso S, Raimondo P, D'Antini D, Mirabella L, Rauseo M, Dambrosio M. Physiological Effects of the Open Lung Approach in Patients with Early, Mild, Diffuse Acute Respiratory Distress Syndrome: An Electrical Impedance Tomography Study. Anesthesiology. 2015 Nov;123(5):1113-21. doi: 10.1097/ALN.0000000000000862. PMID 26397017
- [Background] Scholten EL, Beitler JR, Prisk GK, Malhotra A. Treatment of ARDS With Prone Positioning. Chest. 2017 Jan;151(1):215-224. doi: 10.1016/j.chest.2016.06.032. Epub 2016 Jul 8. PMID 27400909